CLINICAL TRIAL: NCT01770743
Title: A Phase 2, Randomized, Parallel-Group, Active-Controlled, Double-Blind Study to Evaluate the Safety and Immunogenicity of AV7909 for Post-Exposure Prophylaxis of Anthrax Using Three Immunization Schedules and Two Dose Levels in Healthy Adult Volunteers
Brief Title: A Phase 2 Safety and Immunogenicity Study for an Anthrax Vaccine Using 3 Schedules and Two Dose Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EBS.AVA.208 / DMID 11-0055; HHSN272201000035C (Other Grant/Funding Number: National Institute of Allergy and Infectious Diseases)
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Results first posted 2015-02-24 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Anthrax
Keywords: post-exposure prophylaxis; toxin neutralization assay
MeSH Terms: conditions — Anthrax | interventions — Biothrax; Anthrax Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- AV7909 (Day 0 and 14) (Experimental): Route of administration: Intramuscular Dose: 0.5 mL Schedule: Day 0 and Day 14
  Interventions: Biological: AV7909
- AV7909 (Day 0 and 28) (Experimental): Route of administration: Intramuscular Dose: 0.5 mL Schedule: Day 0 and Day 28
  Interventions: Biological: AV7909
- AV7909 (Day 0, 14, and 28) (Experimental): Route of administration: Intramuscular Dose: 0.5 mL Schedule: Day 0, Day 14,and Day 28
  Interventions: Biological: AV7909
- AV7909 Reduced Dose (Experimental): Route of administration: Intramuscular Dose: 0.25 mL Schedule: Day 0, Day 14,and Day 28
  Interventions: Biological: AV7909
- BioThrax (Active Comparator): Route of administration: Intramuscular Dose: 0.5 mL Schedule: Day 0, Day 14,and Day 28
  Interventions: Biological: BioThrax

INTERVENTIONS:
Biological: AV7909 — Anthrax Vaccine Adsorbed plus CPG 7909 Adjuvant
  Other Names: AV7909 Anthrax Vaccine; NuThrax
  Arms: AV7909 (Day 0 and 14); AV7909 (Day 0 and 28); AV7909 (Day 0, 14, and 28); AV7909 Reduced Dose
Biological: BioThrax
  Other Names: Anthrax Vaccine Adsorbed (AVA)
  Arms: BioThrax

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of an anthrax vaccine. The vaccine schedule and dose will also be assessed.

DETAILED DESCRIPTION:
The safety and immunogenicity of AV7909 for post-exposure prophylaxis of anthrax will be evaluated using a randomized, parallel-group, active-controlled, double-blind design with three immunization schedules and two dose levels in healthy adult volunteers. Safety will be assessed by clinical laboratory tests (hematology, serum chemistry, and urinalysis), monitoring of adverse events, vital signs, and physical examinations. Reactogenicity (systemic and injection site reactions) will be assessed by the subjects using subject e-diaries for 7 days after each immunization and by the investigator at in-clinic visits 7 and 14 days after each immunization, and at other visits, if applicable. Immunogenicity will be measured as toxin neutralizing antibody (TNA) response and seroconversion rates.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-50 years old
* Be in good health
* Have access to a computer and the internet so you can complete a diary
* Agree to abstain from sex the first 84 days of the study or practice birth control if you are a woman who is able to get pregnant
* Have not donated blood for the previous 8 weeks

Exclusion Criteria:

* A known anaphylactic response, severe systemic response, or serious hypersensitivity reaction to a prior immunization.
* A history of latex allergy.
* Have received a shot (vaccine), including flu shots, in the past 6 weeks or plan to get a shot for 4 weeks after the last study shot is given.
* Have previously served in the military any time after 1990 or plan to enlist in the military from Screening through Day 84.
* Prior immunization with anthrax vaccine, recombinant protective antigen (rPA) vaccine, or known exposure to anthrax organisms.
* Have participated in anthrax therapeutic or vaccine studies (monoclonal anti-PA or anthrax immune globulins or anthrax vaccines).
* Participation in any investigational study involving use of a pharmacological intervention within 30 days before the Screening visit or planning to participate in a study requiring dosing through the 12-month safety follow-up telephone call.
* Have a known diagnosis of any immunodeficiency disease including but not limited to: acquired immune deficiency syndrome (AIDS), common variable immunodeficiency disease, immunoglobulin A (IgA) deficiency, or hypogammaglobulinemia.
* Past history of significant autoimmune disease such as rheumatoid arthritis, lupus erythematous, psoriasis in the area of vaccinations, or requires immunotherapy, glomerulonephritis, or autoimmune thyroiditis.
* Have received immunosuppressive therapy with cytotoxic drugs or Rituximab within the past 2 years.
* A history of cytotoxic chemotherapy or radiation therapy.
* Chronic (>10 days) daily oral or parenteral corticosteroid therapy in the past 12 months.
* Any lung disease, including reactive airway disease, which requires the daily use of medications.
* A female currently breastfeeding or with a positive pregnancy test.
* A history of drug or alcohol abuse within 12 months prior to Screening, or a positive result on a urine drug screen for cocaine, marijuana, opiates, methamphetamines, benzodiazepines, or oxycodone.
* Any tattoo or other skin condition in the deltoid region on either arm that may obscure the assessment of the injection sites.
* A medical condition that, in the opinion of the PI or designee, could adversely impact the subject's participation or safety or the conduct of the study.
* Any planned elective in-patient surgery during the study period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gurdyal Kalsi, MD, MTOPRA, Principal Investigator — Emergent BioSolutions
Locations (4):
- United States (4):
  - Miami Research Associates, Miami, Florida
  - Costal Carolina Research, Mt. Pleasant, South Carolina
  - Central Texas Allergy and Asthma, New Braunfels, Texas
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 16 January 2013 to 14 November 2013 at 4 medical centers in the United States.
Pre-assignment Details: All 168 enrolled participants who met eligibility criteria were dosed.
Groups:
- BioThrax: Route of administration: Intramuscular Dose: 0.5 mL Schedule: Day 0, Day 14,and Day 28
  BioThrax
Period: Overall Study
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Started | 44 | 34 | 23 | 44 | 23
Treated | 44 | 34 | 23 | 44 | 23
Completed | 42 | 31 | 22 | 42 | 21
Not Completed | 2 | 3 | 1 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 1
Not completed — Sponsor Terminated Subject | 1 | 0 | 0 | 1 | 0
Not completed — Moving Out of State | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax | Total
Number analyzed (Participants) | 44 | 34 | 23 | 44 | 23 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (9.0) | 32.7 (9.7) | 29.7 (10.2) | 32.8 (9.2) | 32.5 (10.4) | 32.5 (9.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 1 | 0 | 1 | 4
  Between 18 and 65 years | 44 | 32 | 22 | 44 | 22 | 164
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 11 | 22 | 11 | 83
  Male | 22 | 17 | 12 | 22 | 12 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 3 | 1 | 3 | 3 | 2 | 12
  White | 40 | 33 | 20 | 40 | 21 | 154
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 4 | 5 | 4 | 29
  Not Hispanic or Latino | 35 | 27 | 19 | 39 | 19 | 139
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 34 | 23 | 44 | 23 | 168

OUTCOME MEASURES:

1. Primary Outcome: Toxin Neutralizing Antibody (TNA) Level at Day 63
Description: Immunogenicity measured by the lower bound (LB) of the 95% confidence intervals (CIs) for the proportion of subjects in each study arm with Day 63 TNA 50% neutralization factor (NF50) values greater than or equal to threshold
Time Frame: Day 63
Population: Per-protocol Population at Day 63 (randomized subjects who did not have any deviation of 1) history of anthrax vaccination; 2) missing or out of window vaccination at Day 14 or 28; 3) incorrect IMP dose at one or more visits; 4) IMP dose associated with a temperature excursion; 5) prohibited medications; or 6) missing Day 63 immunogenicity data).
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Number analyzed (Participants) | 37 | 27 | 18 | 41 | 21
percentage of participants | 56.8 [39.5 to 72.9] | 100 [87.2 to 100] | 100 [81.5 to 100] | 90.2 [76.9 to 97.3] | 52.4 [29.8 to 74.3]

2. Primary Outcome: Incidence of Adverse Events
Description: Incidence of adverse events (including assessment of symptoms, physical exam findings, clinical laboratory tests, and vital signs) from the time of the first immunization on Day 0 through Day 84
Time Frame: From the time of the first immunization on Day 0 through Day 84
Population: Safety Population (subjects who received at least one dose of IMP)
Measure: Number; unit: participants
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Number analyzed (Participants) | 44 | 34 | 23 | 44 | 23
participants | 36 | 26 | 17 | 35 | 15

3. Secondary Outcome: TNA Level at Day 42
Description: Immunogenicity measured by the percentage of subjects in each study arm with Day 42 TNA NF50 values greater than or equal to threshold
Time Frame: Day 42
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Number analyzed (Participants) | 37 | 26 | 18 | 41 | 20
percentage of participants | 86.5 [71.2 to 95.5] | 100 [86.8 to 100] | 94.4 [72.7 to 99.9] | 97.6 [87.1 to 99.9] | 70.0 [45.7 to 88.1]

4. Secondary Outcome: TNA Level at Day 28
Description: Immunogenicity measured by the percentage of subjects with Day 28 TNA NF50 values greater than or equal to threshold
Time Frame: Day 28
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Number analyzed (Participants) | 37 | 27 | 18 | 41 | 21
percentage of participants | 83.8 [68.0 to 93.8] | 11.1 [2.4 to 29.2] | 94.4 [72.7 to 99.9] | 63.4 [46.9 to 77.9] | 47.6 [25.7 to 70.2]

5. Secondary Outcome: TNA Seroconversion Rate
Description: Immunogenicity measured by the percentage of subjects who have seroconverted (defined as a 4-fold increase over Day 0 in TNA NF50 value) at Days 21, 28, 35, 42, 49, 63, and 84
Time Frame: Up to Day 84
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Number analyzed (Participants) | 37 | 27 | 18 | 41 | 21
percentage of participants
  Day 21 | 63.9 [46.2 to 79.2] | 55.6 [35.3 to 74.5] | 77.8 [52.4 to 93.6] | 22.0 [10.6 to 37.6] | 14.3 [3.0 to 36.3]
  Day 28 | 97.3 [85.8 to 99.9] | 40.7 [22.4 to 61.2] | 94.4 [72.7 to 99.9] | 92.7 [80.1 to 98.5] | 57.1 [34.0 to 78.2]
  Day 35 | 97.1 [85.1 to 99.9] | 96.3 [81.0 to 99.9] | 100 [81.5 to 100] | 95.0 [83.1 to 99.4] | 66.7 [41.0 to 86.7]
  Day 42 | 97.3 [85.8 to 99.9] | 100 [86.8 to 100] | 100 [81.5 to 100] | 100 [91.4 to 100] | 95.0 [75.1 to 99.9]
  Day 49 | 91.9 [78.1 to 98.3] | 100 [85.8 to 100] | 100 [81.5 to 100] | 97.6 [87.1 to 99.9] | 95.0 [75.1 to 99.9]
  Day 63 | 86.5 [71.2 to 95.5] | 100 [87.2 to 100] | 100 [81.5 to 100] | 97.6 [87.1 to 99.9] | 85.7 [63.7 to 97.0]
  Day 84 | 75.7 [58.8 to 88.2] | 100 [86.8 to 100] | 100 [81.5 to 100] | 97.4 [86.5 to 99.9] | 63.2 [38.4 to 83.7]

6. Primary Outcome: Incidence of Serious Adverse Events
Description: Incidence of serious adverse events, from the time of the first immunization on Day 0 through the 12-month safety follow-up telephone call following the last scheduled vaccination
Time Frame: From the time of the first immunization on Day 0 through the 12-month safety follow-up telephone call following the last scheduled vaccination
Population: Safety Population (subjects who received at least one dose of IMP)
Measure: Number; unit: participants
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Number analyzed (Participants) | 44 | 34 | 23 | 44 | 23
participants | 2 | 0 | 0 | 0 | 1

7. Primary Outcome: Incidence of Reactogenicity By Severity
Description: Incidence of solicited systemic reactions and solicited injection site reactions each day for 7 days following each vaccination using subject e-diaries by severity.
  Reactions were graded using the following scale (note, for redness and swelling, the diameter [greater of two perpendicular measurements] was assessed by the subject using an injection site measurement tool):
  Grade 0 (Absent): Symptom not present; Grade 1 (Mild): Symptom present but does not interfere with activities of daily living, or affected area (redness, swelling) measures <3 cm; Grade 2 (Moderate): Symptom causes some interference with activities of daily living, or affected area (redness, swelling) measures 3 - 10 cm; Grade 3 (Severe): Symptom prevents activities of daily living or requires treatment, or affected area (redness, swelling) measures > 10 cm.
  For each reaction, subjects are counted once across all vaccinations at the highest reported level of severity.
Time Frame: For 7 days following each vaccination on Days 0, 14, 28
Population: Safety Population (subjects who received at least one dose of IMP)
Measure: Number; unit: participants
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Number analyzed (Participants) | 44 | 34 | 23 | 44 | 23
participants
  Fatigue/Tiredness Grade 1 | 11 | 17 | 14 | 19 | 8
  Fatigue/Tiredness Grade 2 | 6 | 5 | 1 | 2 | 3
  Fatigue/Tiredness Grade 3 | 3 | 0 | 1 | 0 | 0
  Muscle Ache Grade 1 | 25 | 19 | 13 | 27 | 13
  Muscle Ache Grade 2 | 6 | 6 | 7 | 9 | 3
  Muscle Ache Grade 3 | 2 | 0 | 0 | 0 | 0
  Headache Grade 1 | 10 | 15 | 9 | 14 | 8
  Headache Grade 2 | 7 | 3 | 6 | 7 | 1
  Headache Grade 3 | 4 | 0 | 0 | 0 | 0
  Fever Grade 1 | 0 | 0 | 0 | 0 | 0
  Fever Grade 2 | 0 | 1 | 0 | 0 | 0
  Fever Grade 3 | 2 | 0 | 0 | 0 | 0
  Warmth Grade 1 | 17 | 15 | 11 | 14 | 11
  Warmth Grade 2 | 1 | 0 | 2 | 2 | 0
  Warmth Grade 3 | 0 | 0 | 1 | 0 | 0
  Tenderness Grade 1 | 31 | 27 | 17 | 29 | 14
  Tenderness Grade 2 | 11 | 6 | 5 | 9 | 5
  Tenderness Grade 3 | 0 | 0 | 0 | 0 | 0
  Itching Grade 1 | 5 | 3 | 3 | 10 | 5
  Itching Grade 2 | 2 | 0 | 0 | 0 | 0
  Itching Grade 3 | 0 | 0 | 0 | 0 | 0
  Pain Grade 1 | 30 | 29 | 15 | 29 | 14
  Pain Grade 2 | 9 | 2 | 7 | 8 | 6
  Pain Grade 3 | 1 | 0 | 0 | 0 | 0
  Arm Motion Limitation Grade 1 | 21 | 15 | 11 | 17 | 8
  Arm Motion Limitation Grade 2 | 11 | 9 | 7 | 11 | 5
  Arm Motion Limitation Grade 3 | 1 | 0 | 0 | 0 | 0
  Redness Grade 1 | 6 | 5 | 3 | 10 | 8
  Redness Grade 2 | 2 | 1 | 1 | 1 | 0
  Redness Grade 3 | 0 | 0 | 0 | 0 | 0
  Lump Grade 1 | 13 | 6 | 9 | 16 | 10
  Lump Grade 2 | 0 | 0 | 0 | 0 | 0
  Lump Grade 3 | 0 | 0 | 0 | 0 | 0
  Swelling Grade 1 | 12 | 7 | 7 | 14 | 7
  Swelling Grade 2 | 0 | 0 | 2 | 0 | 1
  Swelling Grade 3 | 0 | 0 | 0 | 0 | 0
  Bruise Grade 1 | 4 | 6 | 2 | 8 | 4
  Bruise Grade 2 | 0 | 0 | 0 | 0 | 0
  Bruise Grade 3 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Incidence of Clinical Laborabory Abnormalities
Description: Incidence of clinical laboratory abnormalities throughout the study (up to Day 84).
  Clinical laboratory abnormalities are presented as the total of Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), and Grade 4 (potentially life-threatening) abnormalities according to criteria adapted from the U.S. Department of Health and Human Services, Food and Drug Administration, Center for Biologics Evaluation and Research: Guidance for Industry. Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007). Within each laboratory parameter, subjects are counted once for their most severe occurrence of clinical laboratory abnormality.
Time Frame: From the time of first immunization on Day 0 to Day 84
Population: Safety Population (subjects who received at least one dose of IMP)
Measure: Number; unit: participants
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Number analyzed (Participants) | 44 | 34 | 23 | 44 | 23
participants
  Hemoglobin | 39 | 29 | 20 | 42 | 19
  Leukocytes | 8 | 4 | 3 | 3 | 0
  Neutrophils | 2 | 1 | 1 | 3 | 0
  Lymphocytes | 0 | 1 | 4 | 2 | 0
  Aspartate Aminotransferase | 3 | 2 | 3 | 4 | 1
  Alanine Aminotransferase | 2 | 3 | 1 | 3 | 2
  Glucose | 9 | 7 | 8 | 13 | 2
  Glucose Fasting | 0 | 0 | 1 | 0 | 0
  Bilirubin | 1 | 2 | 1 | 0 | 1
  Blood Urea Nitrogen | 1 | 0 | 1 | 1 | 0
  Urine Glucose | 2 | 1 | 0 | 0 | 1
  Urine Protein | 16 | 10 | 5 | 13 | 6
  Urine Erythrocytes | 11 | 5 | 4 | 7 | 8

9. Primary Outcome: Incidence of Immunologically Significant Adverse Events of Special Interest
Description: Incidence of immunologically significant adverse events of special interest as defined by the Center for Biologics Evaluation and Research from the time of the first immunization on Day 0 through the 12-month safety follow-up telephone call following the last scheduled vaccination
Time Frame: as for outcome 6
Population: Safety Population (subjects who received at least one dose of IMP)
Measure: Number; unit: participants
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Number analyzed (Participants) | 44 | 34 | 23 | 44 | 23
participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of the ICF to the first immunization on Day 0 (AEs recorded only if resulting from a study-related procedure) then through Day 84.
Description: AEs were collected at study visits on Days 0, 7, 14, 21, 28, 35, 42, 49, 63, and 84, and at the early withdrawal visit. The occurrence of SAEs and adverse events of special interest (autoimmune-related) were collected at safety follow-up phone contacts at 6 and 12 months following the last scheduled vaccination.
Arm/Group | AV7909 (Day 0 and 14) | AV7909 (Day 0 and 28) | AV7909 (Day 0, 14, and 28) | AV7909 Reduced Dose | BioThrax
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/34 | 0/23 | 0/44 | 1/23
Other Adverse Events (participants affected / at risk) | 32/44 | 18/34 | 10/23 | 27/44 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AV7909 (Day 0 and 14) (N=44) | AV7909 (Day 0 and 28) (N=34) | AV7909 (Day 0, 14, and 28) (N=23) | AV7909 Reduced Dose (N=44) | BioThrax (N=23)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — cellulitis secondary to animal bite
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — infant of subject experienced one lung underinflated following delivery by precautionary C-section at 36 weeks because of the subject's bicornuate uterus
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AV7909 (Day 0 and 14) (N=44) | AV7909 (Day 0 and 28) (N=34) | AV7909 (Day 0, 14, and 28) (N=23) | AV7909 Reduced Dose (N=44) | BioThrax (N=23)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 5 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 5 (5) | 2 (2) | 7 (8) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/22 (0) | 0/17 (0) | 0/11 (0) | 0/22 (0) | 2/11 (2)
AST increased (Investigations) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 5 (5) | 3 (4) | 2 (2) | 6 (10) | 0 (0)
Blood pressure increased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 1 (2) | 4 (6) | 0 (0) | 1 (1) | 2 (2)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Red blood cells urine positive (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Respiratory rate increased (Investigations) | 6 (14) | 2 (4) | 4 (9) | 10 (13) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A few events collected in e-diary were downgraded (severe to moderate) on verification by the PI but were unable to be corrected in subjects' e-diary data: headache & fatigue/tenderness in 2 subjects each; muscle ache & pain & AML in 1 subject each.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor is responsible for public disclosure of study data. Any proposed publication is subject to review agreed between the Division of Microbiology and Infectious Diseases (DMID) and Emergent; between Emergent and the contract research organizations (CROs)/vendors; and between the CROs and the site Principal Investigator. Data are the property of the sponsor and cannot be published without prior authorization from the sponsor, but data and publication thereof will not be unduly withheld.